CLINICAL TRIAL: NCT03774589
Title: Bilioenteric Anastomosis by Magnetic Compressive Technique: A Prospective, Randomized Controlled Trial
Brief Title: Bilioenteric Anastomosis by Magnetic Compressive Technique
Acronym: BAMCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xi'an Jiaotong University (Other); Northwest Institute for Non-ferrous Metal Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2015-001-1
Record Dates: First submitted 2018-12-12; First posted 2018-12-13 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Pancreatic Cancer; Cholangiocarcinoma; Bile Duct Injury; Choledochal Cyst; Biliary Calculi
Keywords: bilioenteric anastomosis; magnetic compressive technique; morbidity
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Choledochal Cyst; Gallstones

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic Compressive Anastomosis (Experimental): A magnetic device will be used during bilioenteric anastomosis.
  Interventions: Procedure: Magnetic Compressive Anastomosis
- Traditional Manual Anastomosis (Active Comparator): A handsewn technique will be used during bilioenteric anastomosis.
  Interventions: Procedure: Manual Anastomosis

INTERVENTIONS:
Procedure: Magnetic Compressive Anastomosis — The magnetic compressive anastomosis will be used to complete the anastomosis during bilioenteric anastomosis.
  Arms: Magnetic Compressive Anastomosis
Procedure: Manual Anastomosis — A handsewn technique will be used to complete the anastomosis during bilioenteric anastomosis.
  Arms: Traditional Manual Anastomosis

SUMMARY:
The purpose of this study is to determine whether the magnetic compressive anastomosis has a better outcomes than traditional manual anastomosis on bilioenteric anastomosis.

DETAILED DESCRIPTION:
The bilioenteric anastomosis is one of the most common and difficult operations in Hepatobiliary Surgery. The traditional manual anastomosis has become one of the main prognosis factors because of the length of suture time, the difficulty of operation, the high incidence of anastomotic leakage and stricture. Magnetic compressive anastomosis can realize the fast anastomosis, reduce the difficulty, and reduce the incidence of anastomotic leakage and stricture. Currently, the majority of studies of magnetic compressive bilioenteric anastomosis are merely confined within clinical case report and single-center, small sample, retrospective study. This study is a prospective, randomized controlled trial. To evaluate the security, reliability and convince of magnetic compressive bilioenteric anastomosis versus traditional suture method on incidence of anastomotic leakage and stricture between magnetic compressive anastomosis and traditional manual anastomosis among patients who need bilioenteric anastomosis operation. The study is to enroll about 200 patients and divide into Study Group (Group A: Magnetic compressive anastomosis) and Control Group (Group B: traditional manual anastomosis) as 1:1 ratio randomly by stratification factors. The incidence of anastomotic leakage and stricture, length of bilioenteric anastomosis time, value of serum bilirubin, length of discharge time of magnetic device and mean time of hospital stay will be evaluated. The patients will drop out of the study if adverse events happen, active request for dropping out, new-onset severe disease or death. The primary and secondary end point will be observed by regular follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 to 75
* Patients' gender was not limited
* Patients who were well-diagnosed and had the indication for bilioenteric anastomosis.
* Patients whose lifetimes will be longer than 12 months.
* Patients who are willing to join this clinical trial and informed consent form voluntarily.

Exclusion Criteria:

* Woman during pregnancy or lactation or anyone with mental disorder
* The wall of hepatic duct or jejunum was too thick so that the attractive force of magnetic device cannot meet the requirements of compression.
* Any anatomical variation in bile ducts system or the inner diameter is too small so that the magnetic device cannot place in.
* Any foreign body has been implanted in body, such as heart pacemaker.
* Surgical contraindication, including:

Child-Pugh C with hepatic encephalopathy Anyone with heart, lung, kidney dysfunction or other organ dysfunction, and cannot tolerate surgery.Hepatic ducts stone disease, who was diagnosed as Acute Cholangitis of Severe Type, especially complicated with bacteremia or septic shock. End stage disease, complicated with biliary cirrhosis or portal hypertension.Patients with long- term obstructive jaundice, dehydration, electrolyte disturbance or coagulation defects; Patients have the tendency or history of bleeding.

• Any other disease in perioperation periods which needs MRI examination in the next 8 weeks post operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Bilioenteric anastomotic leakage | 1 month post operation
  To compare the incidence of biliary leakage after magnetic or hand-sewn anastomosis

SECONDARY OUTCOMES:
Length of bilioenteric anastomosis time | during operation
  To compare the anastomotic time between magnetic and hand-sewn groups
Time from the date of operation to expel of the magnets. | 1 to 4 weeks postoperation
  To confirm the safe discharge of the magnets
average length of postoperative hospital stay | 3 months
  To compare the length of stay between magnetic and hand-sewn groups
Bilioenteric anastomotic stricture | 1,3,6,12-month post operation
  To compare the long-term outcome between magnetic and hand-sewn groups

CONTACTS AND LOCATIONS:
Overall Officials: Yi Lv, MD,PHD, Principal Investigator — China, Shaanxi First Affiliated Hospital of Xian JiaotongUniversity
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided